CLINICAL TRIAL: NCT00833755
Title: Effect of Ketamine on Opioid-Induced Hyperalgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jianren Mao, MD, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2008P 000879
Record Dates: First submitted 2009-01-29; First posted 2009-02-02 (Estimated); Results first posted 2017-01-16 (Estimated); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Pain; Chronic Pain; Hyperalgesia
Keywords: Pain; Chronic pain; Opioid induced hyperalgesia; Opioid therapy
MeSH Terms: conditions — Pain; Chronic Pain; Hyperalgesia | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Opioid - Ketamine (Active Comparator): This group consists of 16 subjects who have chronic pain conditions treated with an opioid regimen. Subjects were randomized to receive a ketamine treatment during the study. They were given an intravenous infusion of ketamine (0.05mg/kg) diluted in 50 ml normal saline over 30 minutes.
  Interventions: Drug: Ketamine
- Non-opioid - Ketamine (Active Comparator): This group consists of 22 subjects who have chronic pain conditions but were not on an opioid regimen over the last 3 months. Subjects were randomized to receive a ketamine treatment during the study. They were given an intravenous infusion of ketamine (0.05mg/kg) diluted in 50 ml normal saline over 30 minutes.
  Interventions: Drug: Ketamine
- Opioid - Placebos (Placebo Comparator): This group consists of 18 subjects who have chronic pain conditions treated with an opioid regimen. Subjects were randomized to receive a placebo treatment during the study. They were given an intravenous infusion of 50 ml normal saline over 30 minutes.
  Interventions: Drug: Placebos
- Non-opioid - Placebos (Placebo Comparator): This group consists of 23 subjects who have chronic pain conditions but were not on an opioid regimen over the last 3 months. Subjects were randomized to receive a placebo treatment during the study. They were given an intravenous infusion of 50 ml normal saline over 30 minutes.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Ketamine — To compare pain threshold, pain tolerance, and wind up, as measured by QST, before and after a single dose of ketamine infusion under two clinical conditions: chronic pain patients on opioid therapy and chronic pain patients without opioid therapy.
  Other Names: Ketalar
  Arms: Non-opioid - Ketamine; Opioid - Ketamine
Drug: Placebos — To compare pain threshold, pain tolerance, and wind up, as measured by QST, before and after a single dose of ketamine infusion under two clinical conditions: chronic pain patients on opioid therapy and chronic pain patients without opioid therapy.
  Other Names: Saline
  Arms: Non-opioid - Placebos; Opioid - Placebos

SUMMARY:
The purpose of this study is to compare pain threshold, pain tolerance, and wind up, as measured by QST, before and after a single dose of ketamine infusion under two clinical conditions: chronic pain patients on opioid therapy and chronic pain patients without opioid therapy.

DETAILED DESCRIPTION:
We hypothesize that:

1. Chronic pain patients on chronic opioids would have a lower pain threshold and lower pain tolerance when compared to opioid naïve patients (patients with chronic pain with non-opioids treatment)., as measured by QST in a non-affected neutral limb;
2. Chronic pain patients on chronic opioids would have an increased response to painful stimulation, so called "windup" as demonstrated by QST;
3. Both "wind-up" and altered pain threshold and tolerance would be indicative of the presence of opioid-induced hyperalgesia;
4. Intravenous ketamine, an NMDA receptor antagonist, could be used to differentiate between opioid-induced hyperalgesia and opioid tolerance.

ELIGIBILITY:
Inclusion Criteria for Group 1

1. Subject will be between ages 18 to 65 years.
2. Subject has a chronic pain condition for at least three months. This requirement is set in order to avoid the clinical uncertainty of an unstable pain condition and to minimize the study variation. Subjects should have a VAS pain score at 4 or above at the time of study.
3. Subject is on a chronic opioid treatment regimen (e.g., morphine, fentanyl, oxycodone, methadone, hydromorphone, hydrocodone) for at least three months. There should have been no changes in the type and amount of opioid dose for at least one month. Only patients with a minimal daily dose of at least 60 mg morphine equianalgesic dose will be included.

Inclusion Criteria for Group 2

1. Subject who meets the criteria #1 & #2 as listed for Group 1.
2. Subject has not been on an opioid regimen for the last three or more months.

Exclusion Criteria for all groups:

1. Subject has an altered sensation at the skin site of QST (one of upper extremities).
2. Subject has scar tissue or acute injury at the skin site of QST.
3. Subject has neurological disease or a condition causing upper extremities or generalized polyneuropathy, such as diabetic neuropathy, alcoholic neuropathy, AIDS neuropathy, multiple sclerosis, amyotrophic lateral sclerosis, and post-stroke residual neurological deficits.
4. Subject has a diagnosis of renal or liver failure.
5. Subject has a diagnosis of unstable angina, congestive heart failure, cardiac arrythmias or myocardial infarction within 1 year.
6. Subject is allergic to ketamine.
7. Subject had recent therapy that may influence QST results, e.g., neuroablative procedure involving upper extremities within six-months or peripheral neurolytic block involving upper extremities within two-months.
8. Subject has a confirmed diagnosis of and is under the care of a psychiatrist for major depression disorder, eating disorder; alcohol or drug dependence; or attention deficit hyperactivity disorder. Subject has any history of a confirmed diagnosis of bipolar disorder, schizophrenia, anxiety disorder or a psychotic disorder
9. Subject is tested positive on drug urine screening test.
10. Subject is pregnant or breast-feeding.

    -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2008-09; Primary Completion 2013-05 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jianren Mao, M.D., Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luna IE, Kehlet H, Jensen CM, Christiansen TG, Lind T, Stephensen SL, Aasvang EK. The Effect of Preoperative Intra-Articular Methylprednisolone on Pain After TKA: A Randomized Double-Blinded Placebo Controlled Trial in Patients With High-Pain Knee Osteoarthritis and Sensitization. J Pain. 2017 Dec;18(12):1476-1487. doi: 10.1016/j.jpain.2017.07.010. Epub 2017 Aug 24. PMID 28842370
- [Derived] Maher DP, Zhang Y, Ahmed S, Doshi T, Malarick C, Stabach K, Mao J, Chen L. Chronic Opioid Therapy Modifies QST Changes After Ketamine Infusion in Chronic Pain Patients. J Pain. 2017 Dec;18(12):1468-1475. doi: 10.1016/j.jpain.2017.07.008. Epub 2017 Aug 10. PMID 28802882
- See also: MGH Center for Translational Pain Research — http://www.massgeneral.org/translationalpainresearch/

RESULTS

PARTICIPANT FLOW:
Groups:
- Opioid - Ketamine: Subjects who have chronic pain conditions treated with an opioid regimen will be randomized to receive a ketamine treatment during the study.
- Opioid - Placebos: Subjects who have chronic pain conditions treated with an opioid regimen will be randomized to receive a placebo treatment during the study.
- Non-opioid - Ketamine: This group will include subjects who have chronic pain conditions but not on an opioid regimen over the last 3 months. Subjects in this group will be randomized to receive a ketamine treatment.
- Non-opioid - Placebos: This group will include subjects who have chronic pain conditions but not on an opioid regimen over the last 3 months. Subjects in this group will be randomized to receive a placebo treatment.
Period: Overall Study
Arm/Group | Opioid - Ketamine | Opioid - Placebos | Non-opioid - Ketamine | Non-opioid - Placebos
Started | 16 | 18 | 22 | 23
Completed | 12 | 13 | 20 | 17
Not Completed | 4 | 5 | 2 | 6
Not completed — Physician Decision | 4 | 4 | 2 | 6
Not completed — Subject had scheduling issues | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Opioid - Ketamine | Opioid - Placebos | Non-opioid - Ketamine | Non-opioid - Placebos | Total
Number analyzed (Participants) | 16 | 18 | 22 | 23 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 18 | 22 | 23 | 79
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 15 | 13 | 46
  Male | 6 | 10 | 7 | 10 | 33

OUTCOME MEASURES:

1. Primary Outcome: Change in Temperature of Pain Threshold
Description: We measured the change in pain threshold using Quantitative Sensory Testing (QST). QST refers to a set of quantitative testing of individual responses to mechanical, thermal, and/or electrical stimulation. In this study, pain threshold was the thermal stimulation intensity (in°C) first perceived as painful. To measure this, a contact thermode was attached onto the dorsal surface of the forearm. By pressing a computer mouse button, each subject was able to stop stimulation when they first perceived a painful stimulation from the thermode as the temperature increased 1°C/s.
  This test was repeated 3 times and an average temperature was calculated. The temperatures could range from a minimum of 0°C to 53°C.
Time Frame: Baseline at visit 1, post inufsion at visit 1, and at visit 2 which was 1 week after visit 1
Population: Only subjects who experienced pain relief after the infusion were scheduled for visit 2. This is why the overall # of participants analyzed differs from the # of baseline participants.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Opioid - Ketamine | Opioid - Placebos | Non-opioid - Ketamine | Non-opioid - Placebos
Number analyzed (Participants) | 7 | 2 | 4 | 3
Degrees Celsius | -0.02 (0.79) | -0.61 (1.79) | -0.61 (1.15) | -0.77 (1.04)
Statistical Analysis 1: Comparison: Opioid - Ketamine vs Opioid - Placebos vs Non-opioid - Ketamine vs Non-opioid - Placebos; Test type: Superiority or Other; p = 0.274, Kruskal-Wallis

2. Primary Outcome: Change in Temperature of Pain Tolerance
Description: Using QST, we measured the change in pain tolerance which was the maximum thermal stimulation intensity (in °C) tolerable. In this test, the subject was instructed to press the computer mouse to stop stimulation when the thermode reached the maximal tolerable temperature.
  This test was repeated 3 times and an average temperature was calculated. The temperatures could range from a minimum of 0°C to 53°C.
Time Frame: Baseline at visit 1, post inufsion at visit 1, and at visit 2 which was 1 week after visit 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Groups:
- Opioid - Placebo: Subjects who have chronic pain conditions treated with an opioid regimen will be randomized to receive a placebo treatment during the study.
Arm/Group | Opioid - Ketamine | Opioid - Placebo | Non-opioid - Ketamine | Non-opioid - Placebos
Number analyzed (Participants) | 7 | 2 | 4 | 3
Degrees Celsius | -0.06 (1.46) | 0.52 (1.33) | -0.42 (1.95) | -0.19 (1.03)
Statistical Analysis 1: Comparison: Opioid - Ketamine vs Opioid - Placebo vs Non-opioid - Ketamine vs Non-opioid - Placebos; Test type: Superiority or Other; p = 0.552, Kruskal-Wallis

3. Primary Outcome: Change in Duration of Supra-threshold Pain Tolerance
Description: Using QST, we detected the duration (seconds) of tolerance to supra-threshold heat pain stimulation. In this test, subjects were asked to tolerate, as long as he or she could, heat stimulation preset at 47°C for a maximum of 60 seconds. They were given the computer mouse to stop the test if they reached their limit before 60 seconds. If they stopped the test before the 60 seconds, the time that they stopped it was recorded.
  This test was repeated 3 times and an average duration was calculated. The duration could range from a minimum of 0 seconds to a maximum of 60 seconds.
Time Frame: Baseline at visit 1, post inufsion at visit 1, and at visit 2 which was 1 week after visit 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Opioid - Ketamine | Opioid - Placebos | Non-opioid - Ketamine | Non-opioid - Placebos
Number analyzed (Participants) | 7 | 2 | 4 | 3
seconds | -5.22 (9.96) | 13.81 (19.55) | -1.91 (7.32) | -0.39 (13.25)
Statistical Analysis 1: Comparison: Opioid - Ketamine vs Opioid - Placebos vs Non-opioid - Ketamine vs Non-opioid - Placebos; Test type: Superiority or Other; p = 0.004, Kruskal-Wallis

ADVERSE EVENTS:
Groups:
- Opioid - Ketamine; Opioid - Placebos: Subjects who have chronic pain conditions treated with an opioid regimen will be randomized to receive a placebo treatment during the study.
Arm/Group | Opioid - Ketamine | Opioid - Placebos | Non-opioid - Ketamine | Non-opioid - Placebos
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/18 | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 0/16 | 0/18 | 0/22 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No